CLINICAL TRIAL: NCT02530138
Title: The Effect of Synbiotics Supplement on Lipid Profile, Liver Enzymes, Inflammatory Factors and Hepatic Fibrosis in Lean and Normal Weight Patients With Nonalcoholic Fatty Liver
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, associate prof, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 563
Record Dates: First submitted 2015-08-18; First posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Non Alcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Synbiotic (Active Comparator): 2 synbiotic capsules for 28 weeks
  Interventions: Dietary Supplement: synbiotic
- maltodexterin (Placebo Comparator): two capsules per day for 28 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: synbiotic — 2 symbiotics capsules per day for 28 weeks
  Arms: Synbiotic
Dietary Supplement: Placebo — 2 placebo capsules per day for 28 weeks
  Arms: maltodexterin

SUMMARY:
Introduction: Currently, Nonalcoholic Fatty Liver Disease (NAFLD) is the most common liver disease in the world. The only approved treatment for it is lifestyle modification and weight loss; however, there is no evidence for patients with normal or low body mass index (BMI).

The aim of this study is to evaluate the efficacy of symbiotic supplementation in NAFLD patients with normal or low BMI.

Methods and analysis: In this randomized, double-blind, placebo-controlled clinical trial protocol, 21 cases and 21 controls will be individually matched based on age and sex. This 42 patients with NAFLD will be supplemented twice daily for 28 wk with either a synbiotic or a placebo capsule. Both groups will be advised to follow an energy balanced diet and physical activity recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 70 years
* Body Mass Index (BMI) below 25
* Serum alaninaminotransferase more than 1.5 fold of upper limit of normal range
* Sonographic findings compatible with hepatic steatosis (degree 2 or more)

Exclusion Criteria:

* Diabetes
* Taking any kind of antibiotics two weeks before recruitment
* History of alcohol consumption
* pregnancy or lactation
* Professional athletes
* Other liver disease (viral/etc)
* Use of drugs such as calcium channel blockers, high dose synthetic estrogens, methotrexate , amiodarone, steroids, chloroquine, immunosuppressive drugs, lipid-lowering agents, metformin and vitamin E
* A history of Hypertension, Cardiovascular disease, Pulmonary disease, Renal disease & Celiac disease; Cirrhosis
* History of Upper GI surgery / Prior surgical procedures such as jejunoileal or jejunocolic bypass, gastroplasty
* Following program to lose weight in recent 3 mo
* A history of hypothyroidism or Cushing's syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Alaninaminotransferase (ALT) (UL) | 28 weeks
  by biochemical method
hepatic steatosis (cap score) | 28 weeks
  using transient elastography

SECONDARY OUTCOMES:
Body Mass Index (BMI) (kg/m2) | 28 weeks
  using formula

CONTACTS AND LOCATIONS:
Locations (1):
- NNFTRI clinic, Tehran, Tehran Province, Iran